CLINICAL TRIAL: NCT00788424
Title: Study of Topical Application of AS101 for the Treatment of Psoriasis
Brief Title: Topical Application of AS101 for the Treatment of Psoriasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's considerations
Sponsor: BioMAS Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #72REV00
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2008-06

CONDITIONS: Mild to Moderate Psoriasis
Keywords: AS101 Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AS101 Cream (Experimental): Twice daily topical application of AS101 cream on the psoriatic lesions for approx. 12 weeks is expected to clear the treated area.
  Interventions: Drug: AS101 Cream
- Placebo (Experimental): Twice daily topical application on the psoriatic lesions for 8 weeks will serve as control group.
  Interventions: Drug: AS101 Cream

INTERVENTIONS:
Drug: AS101 Cream — 4% AS101 Cream or Placebo cream, twice a day for 12 weeks

SUMMARY:
This protocol relates to a phase II randomized double blind, placebo controlled study of the AS101 topical application for the treatment of mild to moderate Psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient have a diagnosed mild to moderate stable plaque type psoriasis (less than 10% of body skin surface).
2. Patient must be 18-70 years of age.
3. General health must be adequate to allow for compliance with the requirements of this protocol.
4. Patient or his/her legal guardian must sign an informed consent form prior to study participation.
5. Patient must be able and willing to comply with all protocol requirements.

Exclusion Criteria:

1. Patients who are mentally disabled or are otherwise unable to provide fully informed consent.
2. Pregnant or breast-feeding females.
3. Patients with evidence of an infection in the targeted zones.
4. Patients with known sensitivity to any of the drug components.
5. Patients treated by systemic anti psoriatic medications within one month prior to the initial treatment with the AS101, or topical anti psoriatic preparations within two weeks prior to the initial treatment with the AS101.
6. Patient with psoriatic arthritis.
7. Patients taking immunosuppressive drugs.
8. Immunocompromised patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the percentege of patients in which modified PASI (mPASI) score reduction of more than 66% from Baseline whithin 12-week treatment period is achieved | 12 weeks treatment and 3 month follow up

SECONDARY OUTCOMES:
The main secondary endpoints are to evaluate safety, tolerability of topical AS010 treatment and long term remission of psoriasis. | 12 weeks treatment and 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Arie Ingbar, Prof, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel